CLINICAL TRIAL: NCT02246257
Title: Multifactorial Intervention to Prevent Cardiovascular Disease in Patients With Early Rheumatoid Arthritis
Brief Title: Early Rheumatoid Arthritis COR Intervention
Acronym: ERACORI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MD, PhD, Annemarie Lyng Svensson (Other)
Responsible Party: Sponsor-Investigator, MD, PhD, Annemarie Lyng Svensson, MD, PhD, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OdenseUH
Record Dates: First submitted 2014-09-17; First posted 2014-09-22 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis; Cardiovascular Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Cardiovascular Diseases | interventions — Simvastatin; Losartan; Metformin; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Other): In the intervention group all patients will receive statins according to national guidelines. Stepwise introduction of pharmacological therapy targeting 1) hyperlipidaemia, 2) hypertension, 3) hyperglycaemia and 4) microalbuminuria and behaviour modification will be controlled by the project team in an outpatient rheumatology department.
  Hyperlipidaemia: LDL > 2.5 is treated with 40 mg Simvastatin; Hypertension: BT > 140/90 mmHg treated with 100 mg OD Losartan; Diabetes: DM BT > 130/80 mmHg treated with 100 mg OD Losartan; Microalbuminuria: Urinary albumin creatinin ratio > 30 mg treated with 100 mg OD Losartan; Hyperglycaemia: HBA1C > 48 mmol/mol treated with 500 mg increased dose to 2,000 mg in 4 weeks Metformin
  Interventions: Other: Simvastatin; Other: Losartan; Other: Metformin; Other: Outpatient rheumatology department
- Control (Other): In the control group patients will be refered to general practice for pharmacological therapy according to national guidelines targeting 1) hyperlipidaemia, 2) hypertension, 3) hyperglycaemia and 4) microalbuminuria.
  Hyperlipidaemia: LDL > 2.5 is treated with 40 mg Simvastatin; Hypertension: BT > 140/90 mmHg treated with 100 mg OD Losartan; Diabetes: DM BT > 130/80 mmHg treated with 100 mg OD Losartan; Microalbuminuria: Urinary albumin creatinin ratio > 30 mg treated with 100 mg OD Losartan; Hyperglycaemia: HBA1C > 48 mmol/mol treated with 500 mg increased dose to 2,000 mg in 4 weeks Metformin
  Interventions: Other: Simvastatin; Other: Losartan; Other: Metformin; Other: Refered to general practice

INTERVENTIONS:
Other: Simvastatin — LDL > 2.5 is treated with 40 mg
  Other Names: Hyperlipidaemia
Other: Losartan — BT > 140/90 mmHg treated with 50 mg OD
  Other Names: Hypertension
Other: Losartan — DM BT > 130/80 mmHg treated with 50 mg OD
  Other Names: Diabetes
Other: Losartan — Microalbuminuria (urinary albumin creatinin ratio > 30 mg) treated with 100 mg OD
  Other Names: Microalbuminuria
Other: Metformin — HBA1C > 48 mmol/mol treated with 500 mg increased dose to 2,000 mg in 4 weeks
  Other Names: Hyperglycaemia
Other: Outpatient rheumatology department — (4 times yearly)
  Other Names: Intervention
  Arms: Intervention
Other: Refered to general practice
  Other Names: Control
  Arms: Control

SUMMARY:
The primary aim of our present study is to evaluate the effect of a targeted, intensified, multidimensional intervention compared to conventional treatment of modifiable risk factors for CVD in patients with early RA. The primary endpoint, a composite of death from cardiovascular causes, non-fatal MI, non-fatal stroke and re-vascularisation, will be assessed after 5years' follow-up.

DETAILED DESCRIPTION:
The study is a prospective randomised open, blinded endpoint trial with balanced randomisation (1:1) conducted in seven outpatient clinics in Denmark. Follow-up visits for patients in the intervention group are scheduled to occur at baseline and then after 2, 4 and 12 weeks and thereafter every third month for 5 years after randomisation. The control group will be monitored for RA disease activity and comorbidity after 2, 4 weeks, 12 weeks and thereafter following national guidelines for RA. Prevention of CVD risk factors in the control group will be treated in general practice according to national guidelines for diabetes (2011), hypertension (2009) and CVD (2013).

ELIGIBILITY:
Inclusion Criteria:

* RA according to the revised American College of Rheumatology (ACR) 2010 criteria and plasma LDL > 2.5mmol/l.

Exclusion Criteria:

* Pregnancy
* Lactation
* Ongoing/previous DMARD therapy
* Ongoing/previous steorid therapy
* Contraindication to any of the trial drugs
* Current infection with parvovirus B19, hepatitis B, hepatitis C or human immune deficiency virus. Previous report of hospitalisation for myocardial ischaemia defined as follows: a) non-fatal myocardial infarction (MI) defined according to national and international guidelines. b) Acute coronary syndrome (ACS) including acute ischaemic symptoms with possible biomarker changes or elctrocardiographic changes that to not meet the criteria for MI, c) angina pectoris, d) revascularisation (percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-09; Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Time to Major Cardiac Event (death from cardiovascular causes, non-fatal myocardial infarction, non-fatal stroke and cardiac revascularization) | Up to 5 years
  Days from randomization to the first of cardiac event. If no event, censoring occurs at earliest of termination date or efficacy cut-off date of 31 December 2020. Events will be adjudicated by an endpoint committee. Kaplan-Meier estimate of the mean.

SECONDARY OUTCOMES:
Time to Death Due to Any Cause | Up to 5 years
  Days from randomization to death. If no death then censoring occurs at earliest of termination date or efficacy cutoff date of 31 Dec 2020. Kaplan-Meier estimate of the mean
Time to Non-cardiovascular Death | Up to 5 years
  Days from randomization to death from a non-cardiovascular cause. If no event, then censoring occurs at earliest of termination date or efficacy cutoff date of 31 Dec 2020. Events will be adjudicated by an endpoint committee. Kaplan-Meier estimate of the mean
Time to Serious Adverse Event (hospitalizations) | Up to 5 years
  Time from randomization to the first venous thromboembolic event. Kaplan-Meier estimate of the mean
The proportion of patients having a treatment success | 1, 2 and 5 years
  * LDL cholesterol < 2.5 mmol/l
  * HbA1c < 48 mmol/mol (HbA1c < 6.5%),
  * Blood pressure < 140/90 mmHg for non-diabetic patients and < 130/80 mm Hg for diabetic patients and normoalbuminuria (urinary albumin creatinine ratio < 30 mg/g) after 1-year of follow-up this in agreement with present national guidelines, which will be adjusted accordingly to any future changes in the respective national guidelines.
  * Low RA disease activity DAS28-CRP < 3.2 and DAS28-CRP < 2.6 at 12, 24 and 60 months. Furthermore, all to hospitalisations will be adjudicated by the event committee

CONTACTS AND LOCATIONS:
Overall Officials: Torkell J Ellingsen, MD, PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Rheumathology, Frederiksberg and Bispebjerg univeristy Hospital, Frederiksberg, Region of Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Svensson AL, Christensen R, Persson F, Logstrup BB, Giraldi A, Graugaard C, Fredberg U, Blegvad J, Thygesen T, Hansen IM, Colic A, Bagdat D, Ahlquist P, Jensen HS, Horslev-Petersen K, Sheetal E, Christensen TG, Svendsen L, Emmertsen H, Ellingsen T. Multifactorial intervention to prevent cardiovascular disease in patients with early rheumatoid arthritis: protocol for a multicentre randomised controlled trial. BMJ Open. 2016 Apr 20;6(4):e009134. doi: 10.1136/bmjopen-2015-009134. PMID 27098820